CLINICAL TRIAL: NCT00517790
Title: An Open-Label, Randomized, Phase 2 Study of Efficacy and Tolerability of ABT-869 in Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study of ABT-869 in Subjects With Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M06-880; 2007-005245-37 (EudraCT Number)
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-01

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: Refractory; Metastatic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — linifanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABT-869 0.25 mg/kg (Experimental): Approximately half of the subjects were randomized to receive the high dose
  Interventions: Drug: ABT-869 .25 mg/kg
- ABT-869 0.10 mg/kg (Experimental): Approximately half of the subjects were randomized to receive the Low Dose
  Interventions: Drug: ABT-869 0.10 mg/kg

INTERVENTIONS:
Drug: ABT-869 .25 mg/kg — Subjects will take linifanib (ABT-869) based on body weight. Dosing will be determined at baseline and will be based on randomization to either 0.10 mg or 0.25 mg of ABT-869 per kilogram of body weight.
  Arms: ABT-869 0.25 mg/kg
Drug: ABT-869 0.10 mg/kg — Subjects will take linifanib (ABT-869) based on body weight. Dosing will be determined at baseline and will be based on randomization to either 0.10 mg or 0.25 mg of ABT-869 per kilogram of body weight.
  Arms: ABT-869 0.10 mg/kg

SUMMARY:
The purpose of this study is to evaluate the effect of the ABT-869 on the NSCLC subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be histologically or cytologically diagnosed with advanced or metastatic NSCLC
* Subjects must have at least one lesion measurable by CT scan as defined by RECIST
* The measurable lesion may have not received radiation therapy
* Subject has an Eastern Cooperative Oncology Group (ECOG) Performance status of 0-2
* Subject has received at least one prior line of systemic treatment but no more than two treatment regimen(s) for advanced or metastatic NSCLC. In addition, the subject may have received systemic neo-adjuvant or adjuvant chemotherapy for NSCLC
* Adequate organ function

Exclusion Criteria:

* Subject has received targeted VEGF/PDGF TKI (tyrosine kinase inhibitor) therapy. Prior Avastin is allowed.
* Subject has untreated brain or meningeal metastases.
* History of greater than 10% weight loss
* Subject has clinically relevant hemoptysis
* The subject has proteinuria CTC Grade > 1
* The subject currently exhibits symptomatic or persistent, uncontrolled hypertension defined as diastolic blood pressure > 100 mmHg or systolic blood pressure > 150 mmHg. Subjects may be re-screened if blood pressure is shown to be controlled with or without intervention.
* The subject has a documented left ventricular ejection fraction < 50%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-08; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Progression Free Rate (PFR) | Week 16

SECONDARY OUTCOMES:
Objective Response Rate | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Justin Ricker, MD, Study Director — AbbVie
Locations (28):
- United States (18):
  - Site Reference ID/Investigator# 7194, Fountain Valley, California
  - Site Reference ID/Investigator# 5617, Los Angeles, California
  - Site Reference ID/Investigator# 7934, Sacramento, California
  - Site Reference ID/Investigator# 5646, Aurora, Colorado
  - Site Reference ID/Investigator# 6627, Waterbury, Connecticut
  - Site Reference ID/Investigator# 7868, Newark, Delaware
  - Site Reference ID/Investigator# 7616, Port Saint Lucie, Florida
  - Site Reference ID/Investigator# 5648, Chicago, Illinois
  - Site Reference ID/Investigator# 6739, Evanston, Illinois
  - Site Reference ID/Investigator# 8100, Harvey, Illinois
  - Site Reference ID/Investigator# 5269, Indianapolis, Indiana
  - Site Reference ID/Investigator# 6042, St Louis, Missouri
  - Site Reference ID/Investigator# 6680, East Orange, New Jersey
  - Site Reference ID/Investigator# 5603, Voorhees Township, New Jersey
  - Site Reference ID/Investigator# 5652, Buffalo, New York
  - Site Reference ID/Investigator# 6184, Charlotte, North Carolina
  - Site Reference ID/Investigator# 6777, Greensboro, North Carolina
  - Site Reference ID/Investigator# 5650, Memphis, Tennessee
- Canada (3):
  - Site Reference ID/Investigator# 6040, Barrie
  - Site Reference ID/Investigator# 5275, Ottawa
  - Site Reference ID/Investigator# 6572, Toronto
- France (3):
  - Site Reference ID/Investigator# 7756, Marseille
  - Site Reference ID/Investigator# 8068, Toulouse
  - Site Reference ID/Investigator# 8069, Villejuif
- Singapore (2):
  - Site Reference ID/Investigator# 5660, Singapore
  - Site Reference ID/Investigator# 5534, Singapore
- Taiwan (2):
  - Site Reference ID/Investigator# 5663, Taichung
  - Site Reference ID/Investigator# 5640, Taipei

REFERENCES:
- [Derived] Tan EH, Goss GD, Salgia R, Besse B, Gandara DR, Hanna NH, Yang JC, Thertulien R, Wertheim M, Mazieres J, Hensing T, Lee C, Gupta N, Pradhan R, Qian J, Qin Q, Scappaticci FA, Ricker JL, Carlson DM, Soo RA. Phase 2 trial of Linifanib (ABT-869) in patients with advanced non-small cell lung cancer. J Thorac Oncol. 2011 Aug;6(8):1418-25. doi: 10.1097/JTO.0b013e318220c93e. PMID 21597387